CLINICAL TRIAL: NCT01005784
Title: Fixed Versus Flexible GnRH Antagonist Initiation
Brief Title: Fixed Versus Flexible Gonadotropin-releasing Hormone (GnRH) Antagonist Initiation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Prof. Basil Tarlatzis, Medical School, Aristotle University of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHR-3
Record Dates: First submitted 2007-11-13; First posted 2009-11-02 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Subfertility
Keywords: GnRH antagonists
MeSH Terms: conditions — Infertility | interventions — cetrorelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fixed (Active Comparator)
  Interventions: Drug: Cetrorelix (Cetrotide)
- flexible (Experimental)
  Interventions: Drug: Cetrorelix (Cetrotide)

INTERVENTIONS:
Drug: Cetrorelix (Cetrotide) — flexible antagonist administration according to specified criteria
  Other Names: Cetrorelix, Cetrotide, Serono
  Arms: flexible
Drug: Cetrorelix (Cetrotide) — fixed antagonist administration on day 6 of ovarian stimulation
  Other Names: Cetrorelix, Cetrotide, Serono
  Arms: fixed

SUMMARY:
This is a comparison of pregnancy achievement between two GnRH antagonist protocols which differ in the timing of GnRH antagonist initiation.

ELIGIBILITY:
Inclusion Criteria:

* < 39 years of age
* BMI 18.5-29.9
* <= 3 previous IVF cycles

Exclusion Criteria:

* PCOS
* Endometriosis

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2005-06; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Luteinizing hormone rise | 3-14 days (duration of ovarian stimulation)

CONTACTS AND LOCATIONS:
Overall Officials: Efstratios Kolibianakis, Principal Investigator — Unit for Human Reproduction
Locations (1):
- Unit for Human Reproduction, Thessaloniki, Greece

REFERENCES:
- [Derived] Kolibianakis EM, Venetis CA, Kalogeropoulou L, Papanikolaou E, Tarlatzis BC. Fixed versus flexible gonadotropin-releasing hormone antagonist administration in in vitro fertilization: a randomized controlled trial. Fertil Steril. 2011 Feb;95(2):558-62. doi: 10.1016/j.fertnstert.2010.05.052. Epub 2010 Jul 16. PMID 20637457